CLINICAL TRIAL: NCT02210741
Title: Next-generation Sequencing (NGS) of Peripheral Blood Immune Repertoire in Graves' Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201312091RINB
Record Dates: First submitted 2014-08-04; First posted 2014-08-07 (Estimated); Last update posted 2014-08-07 (Estimated); Status verified 2014-08

CONDITIONS: Graves Disease
Keywords: immune repertoire; Graves' disease
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Graves' disease (MIM 27500) is the leading cause of hyperthyroidism worldwide. The prevalence of Graves' disease is quite high (2.7% in women), and there is solid evidence of genetic predisposition. Despite its clinical and scientific significance, Graves' disease is still mysterious in terms of its susceptibility genes or pathophysiological mechanisms. The immune repertoire, being the sum of T and B lymphocytes in a body at any given time, is both a snapshot and a historical record of a person's immune function. Thanks to the power of next-generation sequencing (NGS), massively parallel sequencing of the B cell and T cell receptors suddenly becomes plausible, and opens a door for many creative approaches to study immune related diseases. The ultimate goal of this project is to use both the NGS deep sequencing and immune repertoire experiment to perform Graves' disease sub-group genetic fine mapping, and to identify Graves' disease-specific T cell and B cell receptors. Furthermore, using the immune repertoire approach, investigators want to study the critical epitopes of thyroid auto-antigens, and to delineate the pathophysiological steps in various disease stages and in various sub-groups. Investigators expect to solve the immune repertoire of Graves' disease of different sub-group presentations and at various disease activity stages.

ELIGIBILITY:
Patients with Graves disease

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient from our hospital, National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2014-08; Primary Completion 2024-02 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
B lymphocyte and T lymphocyte receptor profiles of Graves' disease patients | Three years
  "B lymphocyte and T lymphocyte receptor profiles" mean the sequence of the receptors and also the quantity of the lymphocytes with those specific receptor sequences.

CONTACTS AND LOCATIONS:
Overall Officials: Tien-Chun Chang, Principal Investigator — Professor of Department of Internal Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan